CLINICAL TRIAL: NCT02252900
Title: Long-term Clinico-radiological Evolution of Patients With Symptomatic and Asymptomatic Brain Lesions During Infectious Endocarditis
Brief Title: Long-term Clinico-radiological Evolution of Patients With Brain Lesions During Infectious Endocarditis
Acronym: POST-IMAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120901; CRC12019 (Other: APHP)
Record Dates: First submitted 2013-12-19; First posted 2014-09-30 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Infectious Endocarditis
Keywords: Brain damages; MRI; infectious endocarditis
MeSH Terms: conditions — Endocarditis, Subacute Bacterial; Brain Injuries | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cerebral MRI during follow-up of IE (Experimental): All patients will undergo the diagnostic test specific to the study (Magnetic resonance imaging)
  Interventions: Other: Magnetic resonance imaging

INTERVENTIONS:
Other: Magnetic resonance imaging — All patients will undergo the diagnostic test specific to the study

SUMMARY:
Primary objective: To describe the evolution of cerebral lesions in IE patients (number of patients with abnormal cerebral MRI in acute phase of IE and during follow-up).

DETAILED DESCRIPTION:
Introduction:

Infectious endocarditis (IE) is a rare disease (1500 cases per year in France) with a poor prognosis (20 % of mortality). Neurological complications participate in the initial morbimortality but their long-term impact is poorly known. The acute neurological complications are symptomatic in approximately a quarter of patients. Neurological lesions are frequently observed using systematic cerebral imaging. In the IMAGE study, systematic cerebral MRI in 130 patients performed during the acute phase of IE allowed found cerebral lesion in 82 % of the patients and in 79 % of patients without neurological symptoms. The evolution of cerebral lesion, including brain micro-bleedings and their impact prognosis are not known.

Hypothesis: Cerebral lesions detected by MRI during the acute phase of infectious endocarditis may involve and may have an impact on functional prognosis.

Primary objective: To describe the evolution of cerebral lesions in IE patients (comparing the proportion of patients with abnormal cerebral MRI in acute phase of IE and during follow-up).

Secondary objectives:

* To compare frequency of different brain damages in acute phase of IE and during follow-up.
* To analyse the relationship between functional and cognitive status and cerebral lesions.
* To analyse the relationship between initial and follow-up cerebral lesions and initials characteristics (microorganisms, anticoagulation, echocardiographic characteristics, valve replacement surgery, type of valvular substitute, mycotic aneurysm embolization)
* To collect plasma during follow-up of IE
* To compare patient characteristics between patients who accept the functional exploration and those who patient refuse
* To describe oral health and oral condition

ELIGIBILITY:
Inclusion Criteria:

* History of Infective endocarditis treated in Bichat Claude Bernard hospital
* Cerebral MRI performed during the acute phase of endocarditis
* Resident in Metropolitan France
* 18 years old or more

Exclusion Criteria:

* Refusal to participate
* Contra indication to MRI scan
* History of allergy to gadolinium
* Pregnancy or lactating female
* Lack of Social Security or CMU (recipient or beneficiary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportion of patients with abnormal cerebral MRI (ischemic or haemorrhagic lesion, infection and cerebral aneurysm) detected at the initial evaluation during the IE acute phase and at the follow-up visit | 1 day

SECONDARY OUTCOMES:
Rankin scale | 1 day
Karnofsky scale | 1 day
Neuropsychologic tests to assess cognitive, executive, language and memory functions (including MMS, BREF, Trail making test, Wisconsin card sorting test, STROOP) | 1 day
IQCODE | 1 day
SF 36 | 1 day
WhOQOL | 1 day
CES-D scale | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Bernard IUNG, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Bichat - Claude Bernard, Paris, France